CLINICAL TRIAL: NCT02254863
Title: Augmentation of Umbilical Cord Blood Transplantation for Inherited Metabolic Diseases With Intrathecal Administration of Human Umbilical Cord Blood-Derived Oligodendrocyte-Like Cells
Brief Title: UCB Transplant of Inherited Metabolic Diseases With Administration of Intrathecal UCB Derived Oligodendrocyte-Like Cells
Acronym: DUOC-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00050198
Record Dates: First submitted 2014-09-23; First posted 2014-10-02 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Adrenoleukodystrophy; Batten Disease; Mucopolysaccharidosis II; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic; Neimann Pick Disease; Pelizaeus-Merzbacher Disease; Sandhoff Disease; Tay-Sachs Disease; Brain Diseases, Metabolic, Inborn; Alpha-Mannosidosis; Sanfilippo Mucopolysaccharidoses
Keywords: Adrenoleukodystrophy; Batten Disease; Hunter Syndrome; Krabbe; Metachromatic Leukodystrophy; ALD; MLD; PMD
MeSH Terms: conditions — Adrenoleukodystrophy; Neuronal Ceroid-Lipofuscinoses; Mucopolysaccharidosis II; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic; Niemann-Pick Disease, Type A; Pelizaeus-Merzbacher Disease; Sandhoff Disease; Tay-Sachs Disease; Brain Diseases, Metabolic, Inborn; alpha-Mannosidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Intrathecal administration of DUOC-01 (Experimental): Administration of DUOC-01, given intrathecally, between day 26 and 28 post unrelated cord blood transplant
  Interventions: Biological: DUOC-01

INTERVENTIONS:
Biological: DUOC-01 — Intrathecal administration of DUOC-01

SUMMARY:
The primary objective of the study is to determine the safety and feasibility of intrathecal administration of DUOC-01 as an adjunctive therapy in patients with inborn errors of metabolism who have evidence of early demyelinating disease in the central nervous system (CNS) who are undergoing standard treatment with unrelated umbilical cord blood transplantation (UCBT). The secondary objective of the study is to describe the efficacy of UCBT with intrathecal administration of DUOC-01 in these patients.

DETAILED DESCRIPTION:
The inherited metabolic disorders (IMD) are a heterogeneous group of genetic diseases, most of which involve a single gene mutation resulting in an enzyme defect. In the majority of cases, the enzyme defect leads to the accumulation of substrates that are toxic and/or interfere with normal cellular function. Often times, patients may appear normal at birth but during infancy begin to exhibit disease manifestations, frequently including progressive neurological deterioration due to absent or abnormal brain myelination. The ultimate result is death in later infancy or childhood.

Currently, the only effective therapy to halt the neurologic progression of disease is allogeneic hematopoietic stem cell transplantation (HSCT), which serves as a source of permanent cellular ERT.3 However, one barrier to the success of this therapy is delayed engraftment of donor cells in the CNS when administered through the intravenous route, which is associated with ongoing disease progression over 2-4 months before stabilization. The engraftment of donor cells in a patient with an IMD provides a constant source of enzyme replacement, thereby slowing or halting the progression of disease.

This study will evaluate the safety of a potential new treatment for patients with certain IMDs known to benefit from HSCT using allogeneic UCB donor cells. The new intervention, intrathecal administration of UCB-derived oligodendrocyte-like cells (DUOC-01) will serve as an adjunctive therapy to a standard UCB transplant. The goal of this therapy is to accelerate delivery of donor cells to the CNS thereby bridging the gap between systemic transplant and engraftment of cells in the CNS and preventing disease progression. The DUOC-01 cells and cells used for HSCT may be derived from the same UCB donor unit, or a second UCB donor unit will be used to manufacture the DUOC-01 cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be age ≥1 week to ≤21 years.
2. Patients must have one of the following inherited metabolic diseases detected by enzyme or mutation analysis, and confirmed by repeat testing on a separately obtained sample:

   Adrenoleukodystrophy (ALD) Batten Disease Hunter Syndrome (MPS II) Krabbe disease (Globoid Leukodystrophy) Metachromatic Leukodystrophy (MLD) Niemann Pick disease type A or B Pelizaeus-Merzbacher disease (PMD) Sandhoff disease Tay Sachs disease. Alpha Mannosidosis Sanfilippo (MPS III)
3. Patients must have neurologic evidence of their disease, either clinically or via neuroimaging or neurophysiological testing. Examples of evidence of neurologic involvement include, but are not limited to the following:

   * Abnormal EEG, Brainstem Auditory Evoked Response (BAER), and/or Visual Evoked Potentials (VEP).
   * Abnormal brain MRI, ie. increased Loes score (measure of white matter damage, demyelination, and brain atrophy) and/or abnormal corticospinal tracts as assessed by MRI with diffusion tensor imaging (DTI).
   * Three or more of the early clinical markers: problems sleeping, increased activity, behavior difficulties, seizure-like activity, chewing behavior, inappropriate bladder training, inappropriate bowel training.
4. Patients must have adequate organ function as measured by:

   * Renal: Serum creatinine ≤ 2.0 mg/dl
   * Hepatic: Hepatic transaminases (ALT/AST) ≤ 5 x normal, bilirubin ≤ 2.0 mg/dl (except in patients with Gilbert's disease or newborns with physiological or breast milk associated jaundice).
   * Cardiac: Normal cardiac function by echocardiogram or radionuclide scan (shortening fraction or ejection fraction

     * 80% of normal value for age). Patients with acquired or congenital cardiomyopathy may receive melphalan as a substitute for cyclophosphamide.
   * Pulmonary: Pulmonary function tests demonstrating FVC, FEV1, and DLCO ≥ 60% of predicted in patients who can complete the testing. If patient cannot perform PFT's, an O2 sat must be >90% on room air.
5. Patients must have an available, suitably matched, banked UCB unit for transplant.
6. Patients must have a performance status as follows: Lansky ≥ 40%, or Karnofsky ≥ 40%
7. Patients must have a life expectancy of ≥ 6 months.

Exclusion Criteria:

1. Prior organ, tissue, or stem cell transplant within 3 years of study entry.
2. Prior participation in any gene or regenerative cell therapy study.
3. Inability to have an MRI scan or lumbar puncture.
4. Intractable seizures.
5. Chronic aspiration.
6. Bleeding disorder.
7. Evidence of HIV infection or HIV positive serology.
8. Uncontrolled bacterial, viral, or fungal infection at the time of pre-UCBT cytoreduction.
9. Inability to obtain patient's, parent's or legal guardian's consent.
10. Requirement of ventilatory support.
11. Pregnant or breastfeeding.
12. Active concurrent malignancy, or receiving concurrent radiotherapy, immunosuppressive medications, or cytotoxic chemotherapy

Ages: 1 Week to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate for Infusional Toxicity | 24 hours after infusion
  Will monitor for fever, vomiting, neck stiffness, seizures, changes in state of consciousness
Evaluate for Neuro Toxicity | 1 month after infusion
  Perform computerized tomography (CT) scan to evaluate for bleeding, tumor formation, central nervous system generalized infiltration

SECONDARY OUTCOMES:
Efficacy determination | 1-5 years
  Perform standard of care follow-up evaluations to include brain magnetic resonance imaging (MRI) with diffuse tensor imaging (DTI), Electroencephalography (EEG), nerve conduction, brainstem auditory evoked response (BAER), visual evoked potential (VEP) and neurocognitive testing. Bench mark results against historical controls previously transplanted by our institution for the past 20 years.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States